CLINICAL TRIAL: NCT06667271
Title: Clinical Evaluation of Posterior Restorations Made With Direct and Indirect Composites
Brief Title: Clinical Evaluation of Direct and Indirect Composites
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Muhammet Karadaş, Clinical Professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: RTEUDHFMKARADAS004
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Dental Caries
Keywords: Dental caries; Restorative material; Composite resin; Indirect restorarion
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The most commonly used materials in the treatment of decayed teeth are amalgam and composite resins. Because amalgam cannot meet the aesthetic expectations of patients and the rapidly increasing belief that it is toxic, its use has decreased considerably. Although composite resins are primarily used in anterior teeth because they provide aesthetically satisfactory results, they have also become the most preferred material in posterior teeth. This shift is largely due to the significant advancements in their mechanical properties, such as improved strength and durability. Indirect restorations have begun to be used to overcome the disadvantages of resin composites applied with the direct method. Both composite resins and ceramics have given good results for such restorations. However, composite resins have the advantage of being cheaper, more user-friendly, and repairable than ceramics. Laboratory-prepared composite inlays/onlays are more wear-resistant than direct composites, especially in occlusal contact areas. Therefore, they are generally indicated for the restoration of large cavities. Considering the material loss caused by crown restorations and the disadvantages of direct composites in the treatment of teeth with extensive caries, we aimed to treat indirect resin composites that we can apply by making more minimally invasive preparations while supporting the dental tissues.

DETAILED DESCRIPTION:
This study was a double-blind randomized controlled clinical trial involving both evaluators and patients. The research compared indirect restorations with direct restorations. Patients receiving treatment were recalled for follow-ups after one week, six months, and twelve months. Restorations were assessed clinically based on modified FDI criteria, which included marginal discoloration, color match, anatomical form, fracture and retention, marginal adaptation, contact point, postoperative sensitivity, secondary caries, and periodontal response. Qualified clinicians conducted the evaluations using a mirror and probe under reflector light. Additionally, bite-wing radiographs were obtained from patients during the 6-month and 12-month follow-ups to assess the development of secondary caries. Differences between adhesives at each time point were analyzed using Fisher's Exact test, while the effect of time on restorations was evaluated with the Wilcoxon Signed Rank test (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* They have been informed about the study and have agreed to participate.
* They are over 18 years old.
* They do not have any systemic diseases.
* They maintain good general oral health.
* They are not pregnant or breastfeeding.
* The relevant tooth is vital, and the decay is at least 0.5 mm away from the pulp, as confirmed by radiographic findings.
* There is a tooth in contact with the relevant tooth and an antagonist tooth.
* They have agreed to attend follow-up appointments.

Exclusion Criteria:

* After being informed about the study, the participant declined to participate.
* The individual is under 18 years of age.
* The volunteer has a severe systemic disease.
* They have active periodontal or pulp disease.
* They have received endodontic treatment.
* They experience bruxism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The characteristics of the teeth were recorded prior to any restorative procedures. Periapical radiographs were used to assess the status and extent of caries, as well as to identify any potential periodontal or periapical pathologies that might necessitate endodontic treatment. The treated teeth were vital, asymptomatic, and in occlusal contact. Indirect composite restorations were applied to teeth that had caries, old composite or amalgam restorations, secondary caries, or teeth with cuspid loss where the isthmus width exceeded two-thirds of the intercuspal distance.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
World Dental Federation criteria (FDI) | 1 year
  1, Clinically very good; 2, clinically good; 3, clinically sufficient; 4, clinically unsatisfactory; 5, clinically poor

CONTACTS AND LOCATIONS:
Locations (1):
- 53020, Rize, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Incekara MS, Karadas M. Clinical comparison of direct and indirect class II composite restorations: a prospective 12-month follow-up study. BMC Oral Health. 2025 Jul 19;25(1):1217. doi: 10.1186/s12903-025-06604-z. PMID 40684149